CLINICAL TRIAL: NCT03856983
Title: Benefits of Observing Point-light Displays in Postoperative Rehabilitation of the Total Knee Prosthesis.
Acronym: LOARAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A00450-57
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Knee Surgery; Rehabilitation; Point Light Display

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Control group who will do usual rehabilitation.
- Experimental group (Experimental): Experimental group who will do usual rehabilitation and visualization of point-light human actions
  Interventions: Other: Point light display

INTERVENTIONS:
Other: Point light display — Experimental group who will do usual rehabilitation and visualization of point-light human actions
  Arms: Experimental group

SUMMARY:
The LOARAL project concerns patients who have undergone total knee arthroplasty to treat symptomatic osteoarthritis. Patient will be divided into two groups: a control group where patients will do standard rehabilitation and an experimental group where patients will do standard rehabilitation associated with the judgement of point-light display. The aim of this study is to validate the use of point-light display for the Rehabilitation of patients with a totalarthroplasty of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers over 18 years of age who have undergone knee surgery

Exclusion Criteria:

* Any locomotor condition not due to knee surgery
* Uncorrected visual disturbances
* Comorbidity altering locomotion (history of stroke, neurological condition, inflammatory rheumatism)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Compare the evaluation of the point light display relative to conventional rehabilitation | Rehabilitation during 3 weeks
  The time to realize the time up and go test will be assessed at inclusion and at the end of the program.

SECONDARY OUTCOMES:
Compare the evaluation of the point light display on functional recovery | At the end of the program (3 weeks max)
  Test score the time up and go and test score questionnary WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index, Bellamy et al., 1988).
Compare the evaluation of the point light display on the detection and action recognition | At the end of the program (3 weeks max)
  Percentages of correct recognition of actions on the point light display
Compare the evaluation of the point light display on the feeling of self-efficacy personal | At the end of the program (3 weeks max)
  Test score questionnary of self-efficacy personal (Dumont et al., 2000).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Poitiers, France